CLINICAL TRIAL: NCT00585650
Title: Double-blind, Randomized, Placebo-controlled Study of Recombinant Human Tumor Necrosis Factor Receptor (p75) Fusion Protein Etanercept (Enbrel) in Patients With Moderate to Severe Plaque Psoriasis of the Hands and/or Feet
Brief Title: Study of Tumor Necrosis Factor Receptor Fusion Protein Etanercept (Enbrel) in Psoriasis of the Hands and/or Feet
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Kristen Kelly, Professor and Chair of Dermatology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20065092; Amgen Protocol 20060514 (Other: Amgen 20060514)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Psoriasis
Keywords: palmoplantar psoriasis; etanercept; Enbrel
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Etanercept (Enbrel) 50mg twice weekly injections for 12 weeks
  Interventions: Biological: Etanercept
- Placebo Group (Placebo Comparator): Placebo Injections twice weekly for 12 weeks
  Interventions: Other: Placebo injections

INTERVENTIONS:
Biological: Etanercept — Subcutaneous injections 50 mg Etanercept will occur twice weekly over a 12-week treatment period.
  Other Names: Enbrel
  Arms: Treatment Group
Other: Placebo injections — Placebo injections twice weekly for 12 weeks.
  Arms: Placebo Group

SUMMARY:
The purpose of this research study is to see how well (compared to placebo) Enbrel® (etanercept) 50 mg twice a week for 12 weeks affects plaque psoriasis of the hands and/or feet (palmoplantar psoriasis).

DETAILED DESCRIPTION:
This multicenter investigation is a 12 week, double-blind, randomized trial of etanercept, 50 mg twice weekly versus placebo in subjects with palmoplantar psoriasis (PPP). Subjects who meet the eligibility criteria will be randomized to either 50 mg etanercept twice weekly or placebo. Subcutaneous injections will occur twice weekly at approximately the same time of day over the 12-week treatment period. The primary efficacy endpoint will be assessed after 12 weeks of treatment. At the end of the first 12 weeks, all patients (both treatment and placebo arms) will be treated with etanercept 50 mg twice a week (BIW) for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe palmar plantar psoriasis based on physician's global assessment (PGA).
* Between 18 and 70 years of age
* Negative urine pregnancy test at screening and at baseline
* Sexually active men and women of child-bearing potential must agree to use a medically accepted form of contraception (birth control) during the exclusionary medicine wash-out period and throughout the study.
* Ability to self inject study drug or have a designee who can do so
* Capable of understanding and giving written voluntary informed consent

Exclusion Criteria:

* Previous treatment with Enbrel® (etanercept) or similar drugs
* Receipt of investigational drugs or "biologics" within 4 weeks of the screening visit.
* Evidence of skin conditions (e.g. eczema) other than psoriasis that would interfere with evaluations of the study medication.
* Receipt of any biologic medication within the previous 6 months that resulted in a decreased white blood cell count (cells to help fight infections)
* Ultraviolet light treatment (e.g. UVB, PUVA) within one month prior to study drug initiation.
* Receipt of immune-suppressing drugs other than Rheumatrex® (methotrexate) or Soriatane® (acetretin) within 4 weeks prior to the first dose of study drug. Medications you would not be allowed to take during this study include for example, Cytoxan® (cyclosporine), Imuran® (azathioprine), or Sulfazine® (sulfasalazine). If you remain on Rheumatrex® (methotrexate) (≤25 mg/week) or Soriatane® (acitretin) (≤50 mg/day), you must be considered to have inadequate disease control in the opinion of the investigator based on physician's global assessment. You must have been on a stable dose of systemic treatment for at least 1 month prior to the start of the study medication. You will be required to maintain a stable dose of the systemic treatment throughout the study.
* Use of topical steroids in the past 14 days unless they have been used for longer than 14 days and the severity of disease allows entry into study.
* Systemic steroid use (prednisone, etc).
* Prior or concurrent use of Cytoxan® (cyclophosphamide).
* Elevated liver tests; red blood cell count less than normal; decreased platelet count (cells to help with blood clotting); decreased white blood cell count (cells to fight infection); kidney insufficiency
* Any severe adverse event, infection or abnormal laboratory value at the time of the screening visit that would preclude participation in the study
* Presence of a severe infection, less than 30 days prior to the screening visit or between the screening visit and the first dose of study drug
* Pregnant or breast-feeding females.
* Significant concurrent medical diseases including: Uncompensated congestive heart failure (heart is unable to pump as normal): Myocardial infarction (heart attack) within 12 months of screening period; Unstable or stable angina pectoris (chest pains related to your heart); Uncontrolled high blood pressure
* Severe lung disease requiring medical or oxygen therapy
* History of cancer (other than surgically removed skin cancer and in situ cervical cancer) within 5 years of the screening visit
* History of tuberculosis
* Known to be HIV positive
* Rheumatoid arthritis
* Any neurologic demyelinating disease (such as multiple sclerosis or any neurologic disease causing loss of sensation or loss of normal movement) or seizure disorder
* Current or history of psychiatric disease that would interfere with ability to comply with the study protocol or give informed consent.
* History of alcohol or drug abuse.
* Not up-to-date with all immunizations in agreement with the current immunization guidelines
* Significant exposure to the varicella virus (chicken pox)
* Guttate or generalized pustular psoriasis
* Surgery or trauma within a month of baseline considered by the investigator to represent a significant risk or interfere with patient evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald D Weinstein, M.D., Principal Investigator — University of California, Irvine
Locations (3):
- United States (3):
  - UC Irvine Dermatology Clinical Research Center, Irvine, California
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Dermatology Associates, PLLC, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the dermatology clinics.
Groups:
- Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks: Subjects were randomized to receive etanercept 50mg twice weekly injection for 12 weeks. Subjects were then treated for another 12 weeks with etanercept 50 mg twice weekly. An additional follow-up visit performed on week 28.
- Subjects Receiving Placebo for 12 Weeks: Subjects randomized to receive placebo injection twice weekly for 12 weeks. All subjects receiving placebo were then crossed over to etanercept 50 mg twice weekly for another 12 weeks. An additional follow-up visit was performed on week 28.
Period: Overall Study
Arm/Group | Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks | Subjects Receiving Placebo for 12 Weeks
Started | 8 | 12
Completed | 8 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks: Subjects randomized to use etanercept 50mg twice weekly for 12 weeks.
- Subjects Receiving Placebo for 12 Weeks: Subjects randomized to placebo injection twice weekly for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks | Subjects Receiving Placebo for 12 Weeks | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Achieve a 50% Reduction in the Palmoplantar Psoriasis Severity Index at 12 Weeks.
Description: Psoriasis area and severity index (PASI) is the most widely used tool for the measurement of severity of psoriasis. This tool is used to assess the skin lesions of the entire body however, the palmoplantar psoriasis severity index (PPPASI) is a modified form of the the PASI that is assessed for skin lesions of the hands and feet only. The severity is estimated by three clinical signs: erythema induration and desquamation. Severity parameters are measured on a scale of 0 to 4, with 4 being the most severe.
Time Frame: Week 12
Population: Intention to treat
Measure: Number; unit: participants
Groups:
- Subjects Receiving Placebo for the First 12 Weeks: Subjects randomized placebo injection for 12 weeks.
Arm/Group | Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks | Subjects Receiving Placebo for the First 12 Weeks
Number analyzed (Participants) | 8 | 12
participants | 8 | 12

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 28 week period.
Groups:
- Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks: Subjects randomized to use etanercept 50mg twice weekly for 12 weeks. An additional follow-up visit was performed on week 28.
- Subjects Receiving Placebo for 12 Weeks: Subjects randomized placebo injection for 12 weeks. An additional follow-up visit was performed on week 28.
Arm/Group | Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks | Subjects Receiving Placebo for 12 Weeks
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 3/8 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Receiving Etanercept 50 mg Twice Week for 12 Weeks (N=8) | Subjects Receiving Placebo for 12 Weeks (N=12)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No